CLINICAL TRIAL: NCT07312669
Title: ROP Check Premature Infant Outcomes
Brief Title: ROP Check Database Premature Infant Outcomes
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ROPCHECK24
Record Dates: First submitted 2025-11-23; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Retinopathy of Prematurity (ROP)
Keywords: gestational age, birthweight, race, gender
MeSH Terms: conditions — Retinopathy of Prematurity; Birth Weight; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observation of multi-centered care of infants covered by ROP Check cloud-based database is to compare demographic and clinical risk factors to evaluate and improve vision-protecting guidelines.

DETAILED DESCRIPTION:
Infants from multiple academic and community hospital neonatal intensive care units (NICUs) and their covering ophthalmologists had the serial eye examination and treatment data covered by ROP Check® cloud-based database. ROP Check assists neonatologists to implement guideline scheduling of infants according to the American Academy of Pediatrics (AAP). Outcome included progression to Type 1 retinopathy of prematurity (ROP) and treatment details such as intra-vitreal anti-VEGF injection and peripheral ablative laser. demographic data including birthweight, gestational age, gender, race/ethnicity are analyzed to determine risk factors severe ROP. Blindness-preventing guidelines are reviewed, analyzed and evidence-based updates are proposed.

ELIGIBILITY:
Inclusion Criteria:

* NICU infants

Exclusion Criteria:

* Term birth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NICU babies eligible for ROP examination
Sampling Method: Non-Probability Sample
Enrollment: 7070 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ROP treatment: After examination, whether an infant reaching criteria for treatment and what treatment was given. Document the number and the proportion needing treatment. | 2010 through 2022
  Type 1 ROP

CONTACTS AND LOCATIONS:
Locations (1):
- Alaska Children's EYE & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Undecided
Interest level of other parties

REFERENCES:
- [Background] Arnold RW, Jacob J, Matrix Z. Toward Achieving 100% Adherence for Retinopathy of Prematurity Screening Guidelines. J Pediatr Ophthalmol Strabismus. 2017 Nov 1;54(6):356-362. doi: 10.3928/01913913-20170329-04. Epub 2017 Aug 29. PMID 28850643

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: ROP Study protocol with Statistical Analysis Plan (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT07312669/Prot_SAP_000.pdf